CLINICAL TRIAL: NCT00789373
Title: A Phase 3, Double-Blind, Placebo-Controlled Study of Maintenance Pemetrexed Plus Best Supportive Care Versus Best Supportive Care Immediately Following Induction Treatment With Pemetrexed + Cisplatin for Advanced Non-squamous Non-Small Cell Lung Cancer.
Brief Title: A Study of Induction and Maintenance Treatment of Advanced Non-squamous Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12560; H3E-EW-S124 (Other: Eli Lilly and Company); CTRI/2009/091/000113 (Registry Identifier: India)
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Results first posted 2011-07-18 (Estimated); Last update posted 2018-12-14 (Actual); Status verified 2018-02

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- pemetrexed + cisplatin followed by pemetrexed (Experimental): pemetrexed plus cisplatin followed by pemetrexed plus best supportive care
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Other: Best Supportive Care
- pemetrexed + cisplatin followed by placebo (Placebo Comparator): pemetrexed plus cisplatin followed by placebo plus best supportive care
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: Placebo; Other: Best Supportive Care

INTERVENTIONS:
Drug: Pemetrexed — Induction therapy: 500 mg/m^2, intravenous (IV), on Day 1 of each 21-day cycle for 4 cycles
  Other Names: Alimta; LY231514
Drug: Cisplatin — Induction therapy: Cisplatin: 75 mg/m^2, IV, on Day 1 of each 21-day cycle for 4 cycles
Drug: Placebo — Maintenance therapy: Normal saline (0.9% sodium chloride) administered IV on Day 1 every 21-day cycle until progressive disease or treatment discontinuation
  Arms: pemetrexed + cisplatin followed by placebo
Drug: Pemetrexed — Maintenance therapy: 500 mg/m^2, IV, on Day 1 of each 21-day cycle until progressive disease or treatment discontinuation.
  Other Names: Alimta; LY231514
  Arms: pemetrexed + cisplatin followed by pemetrexed
Other: Best Supportive Care — Best Supportive Care is treatment given with the intent to maximize quality of life. Best Supportive Care excludes any treatment in which the goal is to cure or slow the progression of the study disease. Patients will receive Best Supportive Care as judged by their treating physician. Those therapies considered acceptable include, but are not limited to, palliative radiation to extrathoracic structures, antibiotics, analgesics, antiemetics, thoracentesis, pleurodesis, blood transfusions, and/or nutritional support (enteral or parenteral).

SUMMARY:
This study will compare progression-free survival in patients with advanced non-squamous non-small cell lung cancer. Patients who do not progress following 4 cycles of induction treatment with pemetrexed and cisplatin will be randomized 2:1 to receive either maintenance pemetrexed or placebo.

ELIGIBILITY:
Inclusion Criteria for the Induction Phase:

* You must sign an informed consent document for clinical research.
* You must have Stage IIIB or IV nonsquamous Non-Small Cell Lung Cancer.
* You must at least be able to be physically mobile, take care of yourself, and must be up and about and able to perform light activities such as light housework or office work.
* You are allowed to have had prior radiation therapy as long as it was not to more than 25% of the bone marrow and did not include the whole pelvis. Thoracic radiation must be completed more than 30 days before the study. You must be recovered from the toxic effects (except hair loss).
* You must have at least 1 measurable tumor lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST) guidelines or disease that can be evaluated by computed tomography (CT) Scan.
* Your test results assessing the function of your blood forming tissue, kidneys, and liver must be satisfactory.
* You must be 18 years of age or older.
* Women must be sterile, postmenopausal or on contraception and men must be on contraception or sterile (e.g. post-vasectomy).

Exclusion Criteria for the Induction Phase:

* You cannot have squamous cell and/or mixed small cell, non-small cell lung cancer
* You cannot have received other investigational drugs within the last 30 days of entering the trial.
* You cannot have previously completed or withdrawn from this study or any other study investigating pemetrexed.
* You cannot have other serious on-going illnesses including active infections.
* You cannot have a serious cardiac condition, such as a heart attack, angina, or heart disease within 6 months of entering the trial.
* You cannot have had another form of cancer other than superficial basal cell and superficial squamous (skin) cell cancer, or carcinoma in situ of the cervix within the last 5 years. Patients with a history of low-grade (Gleason score less than or equal to 6) localized prostate cancer will be eligible even if diagnosed less than 5 years ago.
* You cannot have known central nervous system (CNS) metastases, other than treated, stable brain metastasis.
* You cannot be receiving nor have received any prior systemic anticancer therapy for lung cancer (including chemotherapy given after surgery in early-stage treatment).
* You cannot have clinically significant third-space fluid collections (e.g. ascites or pleural effusions that cannot be controlled by drainage or other procedures).
* You cannot have received a recent (within 30 days) or are receiving a yellow fever vaccination.
* You are unable to stop taking more than 1.3 grams of aspirin on a daily basis or other non-steroidal anti-inflammatory drugs (NSAIDs).
* You are unable or unwilling to take folic acid, injections of vitamin B12, or corticosteroids.
* You cannot be pregnant or breastfeeding.

Inclusion criteria at Randomization for the Maintenance Phase:

* You must at least be able to be physically mobile, take care of yourself, and must be up and about and able to perform light activities such as light housework or office work.
* You must have documented radiographic evidence of a tumor response of complete response (CR), partial response (PR), or stable disease (SD) according to the Response Evaluation Criteria in Solid Tumors (RECIST) guidelines. Tumor assessment must occur between Cycle 4 (Day 1) of induction therapy and the date of randomization. This response does not have to be confirmed in order for the patient to be randomized to the maintenance phase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 939 (Actual)
Dates: Start 2008-11; Primary Completion 2010-06 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (68):
- Australia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Adelaide, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankston, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wendouree, Victoria
- Belgium (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aalst
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gilly
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liège
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sint-Niklaas
- Finland (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Espoo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Helsinki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampere
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Turku
- France (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Avignon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dijon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Le Mans
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montpellier
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nantes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vandœuvre-lès-Nancy
- Germany (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gerlingen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Großhansdorf
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ulm
- Greece (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Neo Faliro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pátrai
- India (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangalore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bhopal
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madurai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mumbai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Patna
- Italy (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Avellino
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aviano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lido di Camaiore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pisa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Reggio Emilia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Udine
- Netherlands (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ede
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Groningen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Harderwijk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heerlen
- Poland (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- Portugal (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coimbra
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lisbon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vila Franca de Xira
- Romania (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oradea
- Spain (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manresa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sabadell
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zaragoza
- Turkey (Türkiye) (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bornova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sihhiye
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zeytinburnu
- United Kingdom (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aberdeen, Scotland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guildford, Surrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, West Midlands
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newcastle

REFERENCES:
- [Derived] Middleton G, Gridelli C, De Marinis F, Pujol JL, Reck M, Ramlau R, Parente B, Pieters T, Visseren-Grul CM, San Antonio B, John WJ, Zimmermann AH, Chouaki N, Paz-Ares L. Evaluation of changes in renal function in PARAMOUNT: a phase III study of maintenance pemetrexed plus best supportive care versus placebo plus best supportive care after induction treatment with pemetrexed plus cisplatin for advanced nonsquamous non-small-cell lung cancer. Curr Med Res Opin. 2018 May;34(5):865-871. doi: 10.1080/03007995.2018.1439462. Epub 2018 Mar 27. PMID 29424248
- [Derived] Pujol JL, Paz-Ares L, de Marinis F, Dediu M, Thomas M, Bidoli P, Corral J, San Antonio B, Chouaki N, John W, Zimmermann A, Visseren-Grul C, Gridelli C. Long-term and low-grade safety results of a phase III study (PARAMOUNT): maintenance pemetrexed plus best supportive care versus placebo plus best supportive care immediately after induction treatment with pemetrexed plus cisplatin for advanced nonsquamous non-small-cell lung cancer. Clin Lung Cancer. 2014 Nov;15(6):418-25. doi: 10.1016/j.cllc.2014.06.007. Epub 2014 Jun 21. PMID 25104617
- [Derived] Reck M, Paz-Ares LG, de Marinis F, Molinier O, Sahoo TP, Laack E, John W, Zimmermann AH, Visseren-Grul C, Gridelli C. PARAMOUNT: Descriptive subgroup analyses of final overall survival for the phase III study of maintenance pemetrexed versus placebo following induction treatment with pemetrexed plus cisplatin for advanced nonsquamous non-small-cell lung cancer. J Thorac Oncol. 2014 Feb;9(2):205-13. doi: 10.1097/JTO.0000000000000076. PMID 24419418
- [Derived] Paz-Ares LG, de Marinis F, Dediu M, Thomas M, Pujol JL, Bidoli P, Molinier O, Sahoo TP, Laack E, Reck M, Corral J, Melemed S, John W, Chouaki N, Zimmermann AH, Visseren-Grul C, Gridelli C. PARAMOUNT: Final overall survival results of the phase III study of maintenance pemetrexed versus placebo immediately after induction treatment with pemetrexed plus cisplatin for advanced nonsquamous non-small-cell lung cancer. J Clin Oncol. 2013 Aug 10;31(23):2895-902. doi: 10.1200/JCO.2012.47.1102. Epub 2013 Jul 8. PMID 23835707
- [Derived] Zeng X, Peng L, Li J, Chen G, Tan C, Wang S, Wan X, Ouyang L, Zhao Z. Cost-effectiveness of continuation maintenance pemetrexed after cisplatin and pemetrexed chemotherapy for advanced nonsquamous non-small-cell lung cancer: estimates from the perspective of the Chinese health care system. Clin Ther. 2013 Jan;35(1):54-65. doi: 10.1016/j.clinthera.2012.12.013. PMID 23328269
- [Derived] Gridelli C, de Marinis F, Pujol JL, Reck M, Ramlau R, Parente B, Pieters T, Middleton G, Corral J, Winfree K, Melemed S, Zimmermann A, John W, Beyrer J, Chouaki N, Visseren-Grul C, Paz-Ares LG. Safety, resource use, and quality of life in paramount: a phase III study of maintenance pemetrexed versus placebo after induction pemetrexed plus cisplatin for advanced nonsquamous non-small-cell lung cancer. J Thorac Oncol. 2012 Nov;7(11):1713-21. doi: 10.1097/JTO.0b013e318267cf84. PMID 23059776
- [Derived] Paz-Ares L, de Marinis F, Dediu M, Thomas M, Pujol JL, Bidoli P, Molinier O, Sahoo TP, Laack E, Reck M, Corral J, Melemed S, John W, Chouaki N, Zimmermann AH, Visseren-Grul C, Gridelli C. Maintenance therapy with pemetrexed plus best supportive care versus placebo plus best supportive care after induction therapy with pemetrexed plus cisplatin for advanced non-squamous non-small-cell lung cancer (PARAMOUNT): a double-blind, phase 3, randomised controlled trial. Lancet Oncol. 2012 Mar;13(3):247-55. doi: 10.1016/S1470-2045(12)70063-3. Epub 2012 Feb 16. PMID 22341744
- [Derived] Paz-Ares LG, Altug S, Vaury AT, Jaime JC, Russo F, Visseren-Grul C. Treatment rationale and study design for a phase III, double-blind, placebo-controlled study of maintenance pemetrexed plus best supportive care versus best supportive care immediately following induction treatment with pemetrexed plus cisplatin for advanced nonsquamous non-small cell lung cancer. BMC Cancer. 2010 Mar 8;10:85. doi: 10.1186/1471-2407-10-85. PMID 20211022

RESULTS

PARTICIPANT FLOW:
Groups:
- Induction Pemetrexed + Cisplatin: pemetrexed: 500 mg/m^2, intravenous (IV), on Day 1 of each 21-day cycle for 4 cycles.
  cisplatin: 75 mg/m^2, IV, on Day 1 of each 21-day cycle for 4 cycles.
- Pemetrexed + Cisplatin Followed by Maintenance Pemetrexed: Following Induction, received 500 mg/m^2 maintenance pemetrexed, IV, on Day 1 of each 21-day cycle plus Best Supportive Care until progressive disease (PD) or treatment discontinuation.
- Pemetrexed + Cisplatin Followed by Placebo: Following Induction, received placebo (normal saline [0.9% sodium chloride]) administered IV on Day 1 of every 21-day cycle plus Best Supportive Care until PD or treatment discontinuation.
Period: Induction
Arm/Group | Induction Pemetrexed + Cisplatin | Pemetrexed + Cisplatin Followed by Maintenance Pemetrexed | Pemetrexed + Cisplatin Followed by Placebo
Started | 939 | 0 | 0
Completed | 540 (1 patient received maintenance therapy post-induction but was never randomized.) | 0 | 0
Not Completed | 399 | 0 | 0
Not completed — Adverse Event | 64 | 0 | 0
Not completed — Death Due to study disease | 24 | 0 | 0
Not completed — Death due to adverse event | 19 | 0 | 0
Not completed — Death due to toxicity | 11 | 0 | 0
Not completed — Death due to procedure | 1 | 0 | 0
Not completed — Investigator decision | 7 | 0 | 0
Not completed — Protocol entry criteria not met | 9 | 0 | 0
Not completed — Lost to Follow-up | 6 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Progressive Disease | 220 | 0 | 0
Not completed — Withdrawal by Subject | 37 | 0 | 0
Period: Maintenance
Arm/Group | Induction Pemetrexed + Cisplatin | Pemetrexed + Cisplatin Followed by Maintenance Pemetrexed | Pemetrexed + Cisplatin Followed by Placebo
Started | 0 | 359 | 180
Completed | 0 | 0 | 0
Not Completed | 0 | 359 | 180
Not completed — Adverse Event | 0 | 65 | 12
Not completed — Death due to study disease | 0 | 3 | 1
Not completed — Death due to adverse event | 0 | 4 | 1
Not completed — Death due to toxicity | 0 | 1 | 2
Not completed — Investigator Decision | 0 | 4 | 2
Not completed — Protocol entry criteria not met | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — Progressive Disease | 0 | 253 | 152
Not completed — Withdrawal by Subject | 0 | 21 | 8
Not completed — Sponsor Decision | 0 | 0 | 2
Not completed — Participants On-Going at Data Cut-Off | 0 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Induction Pemetrexed + Cisplatin: pemetrexed plus cisplatin
Arm/Group | Induction Pemetrexed + Cisplatin
Number analyzed (Participants) | 939
Age, Continuous [Median (Full Range); unit: years] | 61.3 [24.4 to 83.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 362
  Male | 577
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 59
  African | 7
  Multiple | 2
  Caucasian | 871
Region of Enrollment [Number; unit: participants]
  Portugal | 38
  Greece | 34
  Finland | 18
  Spain | 65
  Turkey | 33
  United Kingdom | 71
  Italy | 175
  India | 54
  France | 106
  Poland | 34
  Belgium | 53
  Romania | 55
  Australia | 26
  Netherlands | 48
  Germany | 126
  Canada | 3
Smoking Status [Number; unit: participants]
  Ever Smoker | 757
  Never Smoker | 175
  Unknown | 7

OUTCOME MEASURES:

1. Primary Outcome: Investigator-assessed Objective Progression-free Survival (PFS)
Description: Investigator-assessed objective PFS was measured from the date of randomization to the first date of objectively determined progressive disease (PD) or death from any cause. For patients not known to have died as of the data cutoff date and who did not have objective PD, PFS was censored at the date of last objective tumor assessment. PD was determined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. PD = 20% increase in sum of longest diameter of target lesions.
Time Frame: Date of randomization to the date of measured PD or date of death from any cause (up to 19.3 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Pemetrexed + Cisplatin Followed by Maintenance Pemetrexed: pemetrexed and cisplatin followed by maintenance pemetrexed plus best supportive care
- Pemetrexed + Cisplatin Followed by Placebo: pemetrexed + cisplatin followed by placebo plus best supportive care
Arm/Group | Pemetrexed + Cisplatin Followed by Maintenance Pemetrexed | Pemetrexed + Cisplatin Followed by Placebo
Number analyzed (Participants) | 359 | 180
months | 4.11 [3.15 to 4.57] | 2.83 [2.60 to 3.12]
Statistical Analysis 1: Comparison: Pemetrexed + Cisplatin Followed by Maintenance Pemetrexed vs Pemetrexed + Cisplatin Followed by Placebo; 900 patients were planned to be enrolled in order to randomize 558 pts to maintenance therapy. This trial was powered for the primary endpoint, PFS (90% power, assuming 238 events with 52% censoring and a PFS Hazard Ratio (HR)=0.65, alpha=0.05). This trial was also powered for a secondary endpoint, OS (93% power, assuming 390 events with 30% censoring and an OS HR=0.70). Alpha was controlled for both a preliminary analysis (alpha=0.0001) and final analysis of OS (alpha=0.0499); Test type: Superiority or Other; p = 0.00006, Log Rank; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.49 to 0.79]

2. Secondary Outcome: Independently-assessed Objective Progression-free Survival (PFS)
Description: To further evaluate the robustness of the PFS analysis, Lilly established an independent review of PFS to assess the potential for investigator bias in the determination of objective PD. PFS was measured from the date of randomization to the first date of objectively determined PD or death. For patients alive as of the data cutoff date and who did not have PD, PFS was censored at the date of the last objective tumor assessment. PD was determined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. PD = 20% increase in sum of longest diameter of target lesions.
Time Frame: Date of randomization to first date of measured PD or date of death from any cause (up to 19.3 months)
Population: Randomized participants with reviewable scan--(316/359 [88%] Maintenance arm and 156/180 [87%] Placebo comparator arm. The majority of unread scans (12.4%) were due to participants not completing 1 cycle of treatment by the data cutoff date (30 June 2010).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Cisplatin Followed by Maintenance Pemetrexed | Pemetrexed + Cisplatin Followed by Placebo
Number analyzed (Participants) | 316 | 156
months | 3.94 [2.96 to 4.24] | 2.60 [2.23 to 2.92]
Statistical Analysis 1: Comparison: Pemetrexed + Cisplatin Followed by Maintenance Pemetrexed vs Pemetrexed + Cisplatin Followed by Placebo; Test type: Superiority or Other; p = 0.0002, Log Rank; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.51 to 0.81]

3. Secondary Outcome: Overall Survival (OS)
Description: OS is the duration from enrollment to death. For patients who are alive, OS is censored at the last contact.
Time Frame: Date of randomization to the date of death from any cause up to 39.5 months
Population: All randomized participants. In the Pemetrexed maintenance arm 103 (28.7%) participants were censored and in the Placebo maintenance arm 39 (21.7%) participants were censored.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Pemetrexed + Cisplatin Followed by Placebo: pemetrexed and cisplatin followed by placebo plus best supportive care
Arm/Group | Pemetrexed + Cisplatin Followed by Maintenance Pemetrexed | Pemetrexed + Cisplatin Followed by Placebo
Number analyzed (Participants) | 359 | 180
months | 13.86 [12.75 to 16.03] | 11.01 [9.95 to 12.52]
Statistical Analysis 1: Comparison: Pemetrexed + Cisplatin Followed by Maintenance Pemetrexed vs Pemetrexed + Cisplatin Followed by Placebo; Type 1 (alpha) error was controlled for the analyses of both PFS and OS in order to maintain an overall two-sided alpha level of 0.05 using a statistical gatekeeping and alpha spending scheme. The unconditional statistical power of the final OS analysis was 93%; Test type: Superiority or Other; p = 0.0195, Log Rank — The predefined alpha for the final analysis of OS is 0.0498 for the unadjusted log-rank test; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.64 to 0.96] — Unadjusted HR from Cox model with treatment as the only cofactor

4. Secondary Outcome: Change From Baseline in the EuroQol Instrument (EQ-5D) Index Score
Description: The EQ-5D is a generic instrument that describes health status in 5 attributes (mobility, self-care, pain/discomfort, anxiety/depression, usual activities) using a three level scale (no problem, some problems, and major problems). These combinations of attributes are converted into a weighted health-state Index Score according to the United Kingdom (UK) population-based algorithm. The possible values for the Index Score range from -0.59 (severe problems in all 5 dimensions) to 1.0 (no problem in any dimension).
Time Frame: Baseline randomization through 30-day post-discontinuation visit (up to 19.3 months)
Population: Participants who were randomized and completed the EQ-5D at baseline and at least once post-baseline. For Cycle 17 and 18, there is no data available for the pemetrexed + cisplatin followed by placebo arm. No participants completed so zero participants were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pemetrexed + Cisplatin Followed by Maintenance Pemetrexed | Pemetrexed + Cisplatin Followed by Placebo
Number analyzed (Participants) | 303 | 153
units on a scale
  Baseline | 0.77 (0.21) | 0.79 (0.18)
  Cycle 1 Day 1: number analyzed (Participants) | 265 | 132
  Cycle 1 Day 1 | 0.01 (0.15) | -0.01 (0.17)
  Cycle 2 Day 1: number analyzed (Participants) | 241 | 129
  Cycle 2 Day 1 | 0.0 (0.19) | 0.01 (0.17)
  Cycle 3 Day 1: number analyzed (Participants) | 160 | 83
  Cycle 3 Day 1 | 0.0 (0.15) | 0.03 (0.17)
  Cycle 4 Day 1: number analyzed (Participants) | 149 | 66
  Cycle 4 Day 1 | -0.01 (0.15) | 0.02 (0.18)
  Cycle 5 Day 1: number analyzed (Participants) | 108 | 48
  Cycle 5 Day 1 | 0.01 (0.16) | 0.01 (0.22)
  Cycle 6 Day 1: number analyzed (Participants) | 98 | 36
  Cycle 6 Day 1 | -0.02 (0.18) | 0.04 (0.14)
  Cycle 7 Day 1: number analyzed (Participants) | 73 | 21
  Cycle 7 Day 1 | 0.01 (0.20) | 0.01 (0.13)
  Cycle 8 Day 1: number analyzed (Participants) | 64 | 18
  Cycle 8 Day 1 | 0.01 (0.18) | 0.05 (0.15)
  Cycle 9 Day 1: number analyzed (Participants) | 48 | 14
  Cycle 9 Day 1 | -0.03 (0.20) | 0.06 (0.18)
  Cycle 10 Day 1: number analyzed (Participants) | 39 | 11
  Cycle 10 Day 1 | 0.0 (0.16) | 0.08 (0.15)
  Cycle 11 Day 1: number analyzed (Participants) | 33 | 8
  Cycle 11 Day 1 | -0.02 (0.19) | 0.04 (0.17)
  Cycle 12 Day 1: number analyzed (Participants) | 28 | 8
  Cycle 12 Day 1 | -0.06 (0.27) | 0.06 (0.16)
  Cycle 13 Day 1: number analyzed (Participants) | 15 | 3
  Cycle 13 Day 1 | -0.01 (0.27) | 0.0 (0.0)
  Cycle 14 Day 1: number analyzed (Participants) | 11 | 4
  Cycle 14 Day 1 | 0.03 (0.26) | 0.03 (0.05)
  Cycle 15 Day 1: number analyzed (Participants) | 12 | 3
  Cycle 15 Day 1 | -0.07 (0.34) | 0.01 (0.02)
  Cycle 16 Day 1: number analyzed (Participants) | 7 | 1
  Cycle 16 Day 1 | -0.01 (0.36) | 0.0 (0.0)
  Cycle 17 Day 1: number analyzed (Participants) | 3 | 0
  Cycle 17 Day 1 | 0.32 (0.43) |
  Cycle 18 Day 1: number analyzed (Participants) | 2 | 0
  Cycle 18 Day 1 | 0.45 (0.52) |
  30 Day Post-Study Visit: number analyzed (Participants) | 82 | 51
  30 Day Post-Study Visit | -0.13 (0.27) | -0.09 (0.26)

5. Secondary Outcome: Change From Baseline in EuroQol Instrument (EQ-5D) Visual Analog Scale (VAS)
Description: Patients indicate their present health state through completion of the VAS. Possible scores range from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: Baseline randomization through 30-day post-discontinuation visit (up to 19.3 months)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pemetrexed + Cisplatin Followed by Maintenance Pemetrexed | Pemetrexed + Cisplatin Followed by Placebo
Number analyzed (Participants) | 300 | 148
units on a scale
  Baseline | 71.1 (16.6) | 71.0 (15.8)
  Cycle 1 Day 1: number analyzed (Participants) | 266 | 126
  Cycle 1 Day 1 | 1.65 (9.86) | 1.42 (10.2)
  Cycle 2 Day 1: number analyzed (Participants) | 239 | 127
  Cycle 2 Day 1 | 1.24 (11.2) | 3.15 (13.0)
  Cycle 3 Day 1: number analyzed (Participants) | 162 | 81
  Cycle 3 Day 1 | 1.82 (10.9) | 4.90 (16.9)
  Cycle 4 Day 1: number analyzed (Participants) | 147 | 65
  Cycle 4 Day 1 | 0.69 (13.1) | 6.15 (16.4)
  Cycle 5 Day 1: number analyzed (Participants) | 107 | 48
  Cycle 5 Day 1 | 1.55 (12.4) | 5.99 (13.1)
  Cycle 6 Day 1: number analyzed (Participants) | 98 | 36
  Cycle 6 Day 1 | 3.01 (12.5) | 5.76 (12.9)
  Cycle 7 Day 1: number analyzed (Participants) | 74 | 21
  Cycle 7 Day 1 | 2.7 (14.5) | 3.98 (10.9)
  Cycle 8 Day 1: number analyzed (Participants) | 64 | 18
  Cycle 8 Day 1 | 4.12 (14.1) | 7.58 (14.8)
  Cycle 9 Day 1: number analyzed (Participants) | 47 | 14
  Cycle 9 Day 1 | 4.19 (14.2) | 7.61 (16.7)
  Cycle 10 Day 1: number analyzed (Participants) | 37 | 11
  Cycle 10 Day 1 | 5.14 (15.1) | 6.23 (18.7)
  Cycle 11 Day 1: number analyzed (Participants) | 33 | 8
  Cycle 11 Day 1 | 2.58 (14.7) | 0.94 (15.4)
  Cycle 12 Day 1: number analyzed (Participants) | 27 | 8
  Cycle 12 Day 1 | 2.11 (16.0) | 4.63 (13.1)
  Cycle 13 Day 1: number analyzed (Participants) | 14 | 4
  Cycle 13 Day 1 | 6.29 (16.4) | 10.0 (3.27)
  Cycle 14 Day 1: number analyzed (Participants) | 11 | 4
  Cycle 14 Day 1 | 3.64 (18.4) | 14.0 (4.55)
  Cycle 15 Day 1: number analyzed (Participants) | 10 | 3
  Cycle 15 Day 1 | 8.40 (12.9) | 12.0 (3.46)
  Cycle 16 Day 1: number analyzed (Participants) | 6 | 1
  Cycle 16 Day 1 | 5.83 (9.99) | 15.0 (0.0)
  Cycle 17 Day 1: number analyzed (Participants) | 3 | 0
  Cycle 17 Day 1 | 15.7 (21.1) |
  Cycle 18 Day 1: number analyzed (Participants) | 2 | 0
  Cycle 18 Day 1 | 5.0 (14.1) |
  30 days post-study: number analyzed (Participants) | 78 | 49
  30 days post-study | -4.77 (17.3) | -3.92 (16.7)

6. Secondary Outcome: Percentage of Participants With Hospitalizations Due to Adverse Events or Requiring Transfusion (Resource Utilization)
Time Frame: Baseline randomization through 30-day post-discontinuation visit (up to 19.3 months)
Population: All randomized participants
Measure: Number; unit: percentage of participants
Arm/Group | Pemetrexed + Cisplatin Followed by Maintenance Pemetrexed | Pemetrexed + Cisplatin Followed by Placebo
Number analyzed (Participants) | 359 | 180
percentage of participants
  Hospitalization due to Drug-related Adverse Event | 8.4 | 3.3
  Transfusions Packed Red Blood Cells | 12.3 | 4.4
  Transfusions Whole Blood | 1.4 | 0.6
  Transfusions Platelets | 1.4 | 0.6
  Transfusions Fresh Frozen Plasma | 0 | 0.6

7. Secondary Outcome: Percentage of Participants With a Non-Serious Adverse Event (AE) During Maintenance Phase
Description: A summary of non-serious AEs is located in the Reported Adverse Event Module.
Time Frame: Baseline randomization through 30-day post-discontinuation visit (up to 49.7 months)
Population: Randomized population with 2% cut-off threshold for inclusion for 19.3 months and 5% for 49.7 months.
Measure: Number; unit: percentage of participants
Groups:
- Pemetrexed Plus Cisplatin Followed by Maintenance Pemetrexed: pemetrexed and cisplatin followed by maintenance pemetrexed plus best supportive care
- Pemetrexed Plus Cisplatin Followed by Placebo: pemetrexed + cisplatin followed by placebo plus best supportive care
Arm/Group | Pemetrexed Plus Cisplatin Followed by Maintenance Pemetrexed | Pemetrexed Plus Cisplatin Followed by Placebo
Number analyzed (Participants) | 359 | 180
percentage of participants
  Non-Serious AEs at 2% Threshold: up to 19.3 Month | 59.9 | 50.6
  Non-Serious AEs at 5% Threshold: up to 49.7 Months | 75.5 | 62.2

8. Secondary Outcome: Percentage of Participants With Serious Adverse Events During Maintenance Phase
Description: A summary of serious adverse events is located in the Reported Adverse Event Module.
Time Frame: Baseline randomization through 30-day post-discontinuation visit (up to 49.7 months)
Population: Randomized population with all serious adverse events included.
Measure: Number; unit: percentage of participants
Arm/Group | Pemetrexed Plus Cisplatin Followed by Maintenance Pemetrexed | Pemetrexed Plus Cisplatin Followed by Placebo
Number analyzed (Participants) | 359 | 180
percentage of participants
  Serious Adverse Events: up to 19.3 Months | 18.9 | 12.2
  Serious Adverse Events: up to 49.7 Months | 26.2 | 20.0

9. Secondary Outcome: Percentage of Participants With Objective Tumor Response (Response Rate) During Maintenance Phase of Study up to Primary Data Cut-Off
Description: Analysis for combined phases was not performed since response was calculated separately for each phase of study. Response using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Complete Response (CR)=disappearance of all target lesions; Partial Response(PR)is at least a 30% decrease in sum of longest diameter of target lesions; Progressive Disease(PD) is at least a 20% increase in sum of longest diameter of target lesions; Stable Disease(SD)=no change or small changes that do not meet the above criteria for CR, PR, or PD.
Time Frame: Baseline to date of measured progressive disease (up to 19.3 months)
Population: All randomized participants
Measure: Number; unit: percentage of participants
Groups:
- Pemetrexed Plus Cisplatin Followed by Maintenance Pemetrexed: pemetrexed and cisplatin followed by maintenance pemetrexed and best supportive care
Arm/Group | Pemetrexed Plus Cisplatin Followed by Maintenance Pemetrexed | Pemetrexed + Cisplatin Followed by Placebo
Number analyzed (Participants) | 359 | 180
percentage of participants | 46.2 | 42.2

10. Secondary Outcome: Percentage of Participants With Independently-Assessed Objective Tumor Response (Response Rate) During Maintenance Phase Up to Primary Data Cut-Off
Description: Response using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Complete Response (CR)=disappearance of all target lesions; Partial Response (PR) is at least a 30% decrease in sum of longest diameter of target lesions; Progressive Disease (PD) is at least a 20% increase in sum of longest diameter of target lesions; Stable Disease (SD)=no change or small changes that do not meet the above criteria for CR, PR, or PD. Response Rate = (CR+PR)/Participants in Arm*100. Disease Control Rate=(CR+PR+SD)/Number of Participants in Arm*100.
Time Frame: Date of randomization to date of measured PD (up to 19.3 months)
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed + Cisplatin Followed by Maintenance Pemetrexed | Pemetrexed + Cisplatin Followed by Placebo
Number analyzed (Participants) | 359 | 180
percentage of participants
  Response Rate | 46.2 [41.0 to 51.6] | 42.2 [34.9 to 49.8]
  Disease Control Rate | 98.1 [96.0 to 99.2] | 94.4 [90.0 to 97.3]

ADVERSE EVENTS:
Time Frame: From start of study up to approximately 108 months
Arm/Group | Induction Pemetrexed + Cisplatin | Pemetrexed + Cisplatin Followed by Maintenance Pemetrexed | Pemetrexed + Cisplatin Followed by Placebo
Serious Adverse Events (participants affected / at risk) | 257/939 | 94/359 | 36/180
Other Adverse Events (participants affected / at risk) | 759/939 | 287/359 | 117/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Induction Pemetrexed + Cisplatin (N=939) | Pemetrexed + Cisplatin Followed by Maintenance Pemetrexed (N=359) | Pemetrexed + Cisplatin Followed by Placebo (N=180)
Anaemia (Blood and lymphatic system disorders) | 13 (30) | 11 (21) | 1 (1)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 12 (13) | 6 (6) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 3 (3) | 2 (3) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 8 (9) | 6 (8) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (9) | 5 (8) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (3) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (4) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (3) | 0 (0) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 1 (5) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 3 (3) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
Diastolic dysfunction (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0) | 1 (2)
Pericarditis (Cardiac disorders) | 1 (6) | 2 (5) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (14) | 0 (0)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (6) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (11) | 3 (4) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 2 (6) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (8) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 7 (9) | 3 (3) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 4 (6) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (3) | 1 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 3 (6) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 24 (41) | 2 (5) | 1 (1)
Neutropenic colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 29 (36) | 3 (3) | 1 (1)
Asthenia (General disorders) | 5 (9) | 2 (4) | 0 (0)
Chest pain (General disorders) | 7 (17) | 3 (17) | 0 (0)
Death (General disorders) | 5 (5) | 1 (1) | 0 (0)
Fatigue (General disorders) | 7 (22) | 3 (4) | 1 (3)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 7 (10) | 1 (2) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (3) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (3) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 10 (13) | 4 (5) | 2 (2)
Sudden death (General disorders) | 0 (0) | 1 (1) | 1 (1)
Thrombosis in device (General disorders) | 0 (0) | 0 (0) | 1 (10)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (2) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 2 (5) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 3 (7) | 0 (0)
Device related infection (Infections and infestations) | 2 (4) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 3 (10) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 1 (2) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (1) | 1 (2) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 3 (3) | 2 (3) | 1 (1)
Lung abscess (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Lung infection pseudomonal (Infections and infestations) | 1 (3) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 17 (25) | 5 (8) | 3 (3)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (2) | 2 (3) | 0 (0)
Rotavirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Scrotal abscess (Infections and infestations) | 0/577 (0) | 0/201 (0) | 1/112 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (2) | 0 (0) | 1 (3)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (3) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Fracture displacement (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (6)
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Venous injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Biopsy pleura (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine decreased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Blood creatinine increased (Investigations) | 3 (4) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 2 (3) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (2) | 1 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 11 (12) | 1 (2) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (3) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (4) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercreatininaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (5) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 1 (2) | 4 (8)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (9) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (4) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (36) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (6) | 0 (0) | 1 (5)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (7) | 0 (0)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 0 (0)
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (11) | 0 (0) | 0 (0)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 4 (9) | 1 (2) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 6 (9) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 4 (6) | 2 (4) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Facial paresis (Nervous system disorders) | 0 (0) | 1 (4) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 5 (19) | 0 (0)
Hemiplegia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (8) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0)
Paraplegia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Pyramidal tract syndrome (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 1 (2)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1/362 (1) | 0/158 (0) | 0/68 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1/362 (2) | 0/158 (0) | 0/68 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (3) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (2) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (3) | 0 (0) | 0 (0)
Bladder diverticulum (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Incontinence (Renal and urinary disorders) | 1 (6) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 5 (7) | 4 (7) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 7 (9) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 2 (4) | 0 (0) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 1/577 (3) | 0/201 (0) | 0/112 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 1 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 (26) | 6 (12) | 3 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11 (28) | 3 (3) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 28 (63) | 3 (14) | 3 (7)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (6) | 0 (0) | 0 (0)
Catheter removal (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Arterial thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Arterial thrombosis limb (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 4 (6) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (6) | 0 (0) | 0 (0)
Iliac artery thrombosis (Vascular disorders) | 0 (0) | 1 (11) | 0 (0)
Ischaemic limb pain (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Jugular vein distension (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Superior vena caval occlusion (Vascular disorders) | 0 (0) | 1 (3) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction Pemetrexed + Cisplatin (N=939) | Pemetrexed + Cisplatin Followed by Maintenance Pemetrexed (N=359) | Pemetrexed + Cisplatin Followed by Placebo (N=180)
Anaemia (Blood and lymphatic system disorders) | 152 (600) | 76 (295) | 5 (11)
Neutropenia (Blood and lymphatic system disorders) | 158 (340) | 38 (100) | 3 (4)
Constipation (Gastrointestinal disorders) | 131 (339) | 23 (110) | 14 (47)
Diarrhoea (Gastrointestinal disorders) | 114 (175) | 28 (44) | 7 (16)
Nausea (Gastrointestinal disorders) | 362 (932) | 69 (286) | 8 (15)
Vomiting (Gastrointestinal disorders) | 210 (366) | 42 (78) | 9 (14)
Asthenia (General disorders) | 141 (494) | 51 (325) | 8 (16)
Chest pain (General disorders) | 44 (139) | 18 (77) | 6 (13)
Fatigue (General disorders) | 181 (743) | 55 (316) | 16 (61)
Mucosal inflammation (General disorders) | 50 (83) | 21 (50) | 5 (9)
Oedema peripheral (General disorders) | 42 (168) | 45 (314) | 5 (18)
Pyrexia (General disorders) | 46 (63) | 38 (65) | 7 (7)
Decreased appetite (Metabolism and nutrition disorders) | 119 (316) | 32 (91) | 6 (21)
Back pain (Musculoskeletal and connective tissue disorders) | 31 (127) | 23 (155) | 7 (15)
Dizziness (Nervous system disorders) | 30 (76) | 18 (55) | 3 (14)
Paraesthesia (Nervous system disorders) | 17 (76) | 17 (118) | 13 (36)
Cough (Respiratory, thoracic and mediastinal disorders) | 67 (250) | 29 (79) | 11 (26)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 73 (235) | 43 (201) | 17 (54)
Rash (Skin and subcutaneous tissue disorders) | 48 (90) | 15 (65) | 9 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days